CLINICAL TRIAL: NCT03173690
Title: Medicines Reconciliation at an Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: Hospital Pharmacy Enterprise, South Eastern Norway (Other)
Responsible Party: Principal Investigator, Silje Engdal Ørnes, Clinical pharmacist, Ph.d, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-186
Record Dates: First submitted 2017-05-22; First posted 2017-06-02 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Medicines Reconciliation; Intensive Care Unit

STUDY DESIGN:
Intervention Model Description: The included patients are randomized to either intervention or control group. The intervention group receives medicines reconciliation at the intensive care unit. The control group receive standard pharmaceutical care, which now does not include medicines reconciliation. After the patients are transferred to care at the ward, medicines reconciliation is performed for all patients.
Who Masked: Care Provider
Masking Description: The care provider performing medicines reconciliation at ward is semimasked. The masking might be broken if the patients tells if he/she has been interviewed earlier in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive medication reconciliation at the ICU, pluss medication reconciliation at the ward
  Interventions: Other: Medication reconciliation at the ICU; Other: Medication Reconciliation at the Ward
- Control group (Other): No intervention at the ICU, medication reconciliation at the ward
  Interventions: Other: Medication Reconciliation at the Ward

INTERVENTIONS:
Other: Medication reconciliation at the ICU — Medication reconciliation performed according to Integrated Medicines Management model
  Arms: Intervention group
Other: Medication Reconciliation at the Ward — Medication reconciliation performed according to Integrated Medicines Management model

SUMMARY:
This study evaluates the effect of performing medicines reconciliation on patients admitted to an intensive care unit. Half of the patients will receive a medicines reconciliation at the intensive care unit. The other half will not. All included patients will receive medicines reconciliation after transfer to the ward.

DETAILED DESCRIPTION:
Transfer of patients from one level of care to another is known to increase the risk of medication errors. Medication reconciliation is an accepted intervention to increase the knowledge on the patients medication use, thus reducing the risk of avoidable medication errors. For patients in the intensive care unit treatment of the imminent threat is obviously the most important. Nevertheless, knowledge about previous medications are important.

ELIGIBILITY:
Inclusion Criteria:

* belonging to the hospitals intake area
* written informed concent by the patient or his/her next to kin

Exclusion Criteria:

* Patients without next to kin
* Not Norwegian speaking, in need of a translator
* medication reconciliation performed earlier
* Patients with Guillain-Barre or Myasthenia Gravis, due to long expectancy of stay
* Short life expectancy, decided in cooperation with the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one discrepancy between medications listed on hospital chart and medications used at home before hospital admittance | Medicines reconciliation is performed at randomisation and within 48 hours after transmission to the ward, assessed up to 28 days after randomisation
  Medications listed on the medication chart were recorded on a predefined form, this included information on dosage form, strength, dosage and administration time for each drug. The pharmacist performed medicines reconciliation either by interviewing the patient or by gathering information from other sources as the patient's general practitioner, next-to-kin or if relevant nursing home. Any deviations between the information from the medication chart and information obtained during medicines reconciliation was defined as a discrepancy.

SECONDARY OUTCOMES:
Retrospective evaluation on the clinical relevance of the observed medical discrepancies | Retrospectively, based on the information gathered from the day of randomisation up until 28 days after randomisation
  One clinical pharmacist and one senior geriatrician retrospectively asses the potential clinical relevance of the registered discrepancies. The expert panel use the following information for each patient when assessing the clinical relevance: medication list before and after reconciliation, age, gender, reason for hospitalisation, former and current diseases and the level of care before admission

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Oernes, PhD, Principal Investigator — Hospital Pharmacy Enterprise, South Eastern Norway
Locations (1):
- Akershus university Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No